CLINICAL TRIAL: NCT00060515
Title: An Open-Label Dose-Escalation Phase I Study to Asses the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RG2133 (2',3',5'-Tri-O-Acetyluridine) in the Treatment of Inherited Mitochondrial Diseases
Brief Title: RG2133 (2',3',5'-Tri-O-Acetyluridine) in Mitochondrial Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Repligen Corporation (Industry)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: RG2133-01
Record Dates: First submitted 2003-05-07; First posted 2003-05-08 (Estimated); Last update posted 2005-08-05 (Estimated); Status verified 2005-08

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases | interventions — uridine triacetate

INTERVENTIONS:
Drug: RG2133 (2',3',5'-tri-O-acetyluridine)

SUMMARY:
The objective of the study is to determine the safety and tolerability of RG2133 in patients with Mitochondrial Disease.

ELIGIBILITY:
Mitochondrial Disease

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12